CLINICAL TRIAL: NCT07293195
Title: Adjunctive Effects of Heat Versus Contrast Therapy With Otago Exercises on Pain, Swelling, Range of Motion and Functional Limitations in Patients With Patellofemoral Pain Syndrome
Brief Title: Adjunctive Effects of Heat vs Contrast Therapy With Otago Exercises on Patellofemoral Pain Syndrome
Acronym: PFPS OEP CT HT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Principal Investigator, Umber Nawaz, Assistant Professor, Lahore University of Biological and Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LCPT/DPT/ERB/31; U1111-1332-0257 (Registry Identifier: WHO- Universal Trial Number)
Record Dates: First submitted 2025-12-06; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral pain syndrome(PFPS), Heat therapy(HT), Contrast therapy(CT),Otago exercise program(OEP)
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Heat therapy with Otago exercises (Experimental): 1. Heat Therapy:
     * Frequency: 3 sessions/week for 4 weeks
     * Intensity: Mild to moderate heat (40°C)
     * Time: 15 minutes/session
     * Type: Passive superficial heat via electrical hot pack
  2. Otago Exercise Program:
     * Frequency: 3 sessions/week supervised + daily home exercise for 4 weeks
     * Intensity: Progressively increasing strength and balance
     * Time: 30 minutes/session (includes warm-up and cool-down)
     * Type: Functional, strength, and balance exercises for lower limbs
  3. Routine Physical Therapy (Medial Patellar Mobilization):
     * Frequency: 3 sessions/week for 4 weeks
     * Intensity: Gentle grade I/II mobilization
     * Time: 3 sets of 10 repetitions
     * Type: Passive sustained medial glides of patella
  Interventions: Other: Heat therapy+Otago exercise program; Other: Contrast therapy+ Otago exercise program
- Active Experimental Group: Contrast therapy with Otago exercises (Active Comparator): 1. Contrast Therapy:
     * Frequency: 3 sessions/week for 4 weeks
     * Intensity: Heat (38-40°C) and cold (12-14°C)
     * Time: 15 minutes/session (4 min heat + 1 min cold cycles)
     * Type: Alternating hot/cold packs
  2. Otago Exercise Program:
     * Frequency: 3 sessions/week supervised + daily home exercise for 4 weeks
     * Intensity: Progressively increasing strength and balance
     * Time: 30 minutes/session (includes warm-up and cool-down)
     * Type: Functional, strength, and balance exercises for lower limbs
  3. Routine Physical Therapy (Medial Patellar Mobilization):
     * Frequency: 3 sessions/week for 4 weeks
     * Intensity: Gentle grade I/II mobilization
     * Time: 3 sets of 10 repetitions
     * Type: Passive sustained medial glides of patella
  Interventions: Other: Heat therapy+Otago exercise program

INTERVENTIONS:
Other: Heat therapy+Otago exercise program — Heat therapy is a non-surgical technique being recognized for its application in knee pain management. HT enhances blood flow, alleviates pain, and aids tissue repair. It have been effective in knee osteoarthritis but have yet to be fully explored for the treatment of PFPS.
  Other Names: Hot pack; Electrical Hot pack
Other: Contrast therapy+ Otago exercise program — Contrast therapy (CT), a commonly used thermal treatment, is gaining attention as a non-invasive option for managing knee pain. By alternating between heat and cold, CT helps stimulate circulation, reduce swelling, and ease joint stiffness. While it has shown benefits in other knee conditions, its potential role in treating patellofemoral pain syndrome (PFPS) is still not well established.
  Arms: Experimental Group: Heat therapy with Otago exercises

SUMMARY:
The goal of this clinical trial is to determine the adjunctive effects of heat therapy and contrast therapy when combined with the Otago exercise program in individuals with patellofemoral pain syndrome aged 18 to 40 years. The study aims to assess whether these interventions can help reduce pain and swelling, improve knee range of motion, and decrease functional limitations associated with patellofemoral pain syndrome. Researchers will compare two groups one receiving heat therapy with the Otago exercise program and the other receiving contrast therapy with the Otago exercise program to see which approach provides greater improvement in outcomes. Participants will undergo regular supervised sessions that include the assigned thermal therapy and a structured set of Otago exercises targeting lower limb strength, balance, and mobility.

ELIGIBILITY:
Inclusion Criteria:

Participants having age group between 18 and 40 years with anterior, retropatellar, or peripatellar pain with at least severity of 3/10 on the numerical pain rating scale.

Participants who have reported anterior knee pain for at least three months during at least two of the following activities: seating for prolonged periods of time; ascending and descending stairs; squatting; running and jumping, or have had experienced crepitus (popping, or crackling) while walking or running, pain on palpation, insidious pain lasting at least two months.

Positive patellar compression and Grind tests.

Clinical evidence of lateral patellar tracking, given its established role in patellofemoral joint dysfunction.

Pain produced by at least two of the following four tests: (i) isometric muscle contraction with a mild bent knee, (ii) patellofemoral joint line palpation, (iii) compression of patella against the femur and (iv) active resisted knee extension were enrolled in the study.

Exclusion Criteria:

Pain lasting less than three months, previous knee operations, meniscal lesions, patellar instability (subluxation/dislocation), clinical evidence of tendinopathy or ligamentous injury, fractures or dislocations involving the pelvis, spinal surgical history, osteoporosis, pregnancy, neurological diseases or radiological findings of chondromalacia beyond grade 2 on MRI, ultrasound, or X-ray.

Recent participation in lower-limb rehabilitation or structured training within six weeks, or prior diagnoses of rheumatoid arthritis, gout, or other rheumatic knee disorders.

Use of NSAIDs in the preceding four weeks, prior history of cancer, infection, psychiatric conditions, cognitive impairment, autoimmune pathology, or neurological dysfunction likely to interfere with walking ability.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-05-24 (Estimated); Study Completion 2026-05-24 (Estimated)

PRIMARY OUTCOMES:
Swelling | 4 Weeks
  Swelling, also known as edema, is the enlargement of body tissues due to fluid accumulation. It can occur in various parts of the body, such as the hands, feet, ankles, or even internally within organs. Swelling is often a symptom of an underlying condition, including injuries, infections, or medical conditions like heart or kidney problems. Measured by an in elastic tape (Girth measurement)
Pain Intensity | 4 Weeks
  The International Association for the Study of Pain (IASP) 1979 has described Pain as a feeling of discomfort and emotion resulting from actual or potential harm to body tissues. It is a core subjective occurrence, shaped over time by childhood incidents of harm or emotional trauma. From a physiological perspective, pain is triggered by stimuli that pose a risk of tissue injury. Hence, pain is perceived as a conscious and individualized experience with tissue damage potential harm to bodily structures. Assessed by using the NPRS scale.
Range Of Motion | 4 Weeks
  Assessing joint range of motion (ROM) is frequently employed in physiotherapy especially in outpatient orthopedic departments and primary care facilities. Core objectives of physical therapists is to help patients recover their joint flexibility, build strength, and return to normal physical functioning. Assessing range of motion is fundamental for detecting limitations in movement and serves as an essential tool for evaluating progress over time. Measured by Universal goniometer.

SECONDARY OUTCOMES:
Functional limtations | 4 Weeks
  Functional limitation is defined as a loss of functional capability in performing routine mental or physical tasks needed for independent living, without any influence from environmental factors. The Oxford Knee Score (OKS) given by Dawson et al. in 1998 assesses knee pain severity and functional capacity using a scoring system from 0 (most severe impairment) to 48 (full function and no pain).

IPD SHARING:
Plan to Share IPD: Yes
Will be shared after research publication
Supporting Information: Study Protocol, CSR
Time Frame: 6 months
Access Criteria: Researcher, Layman,